CLINICAL TRIAL: NCT05567406
Title: A Phase 2, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of Belumosudil in Black or African American, American Indian or Alaska Native, and Native Hawaiian or Other Pacific Islander Participants With Chronic Graft Versus Host Disease (cGVHD) After At Least 2 Prior Lines of Systemic Therapy
Brief Title: Safety and Efficacy of Oral Belumosudil in Black or African American, American Indian or Alaska Native, and Native Hawaiian or Other Pacific Islander Male and Female Participants Aged 12 Years and Above With Chronic Graft Versus Host Disease (cGVHD) After At Least 2 Prior Lines of Systemic Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFY17661; U1111-1277-6715 (Registry Identifier: ICTRP); KD025-218 (Other: Sanofi Identifier)
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; KD025

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belumosudil (Experimental): Participants will receive belumosudil orally, once daily (QD) or twice daily (BID) if they are taking strong CYP3A4 inducers or proton pump inhibitors.
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Pharmaceutical form: Tablet; Route of administration: Oral
  Other Names: KD025; SAR445761; Rezurock

SUMMARY:
The purpose of this study is to measure safety and efficacy of oral belumosudil in Black or African American, American Indian or Alaska Native, and Native Hawaiian or Other Pacific Islander male and female participants with cGVHD who have previously been treated with at least 2 prior lines of systemic therapy aged 12 years and above.

The duration of participants participation will be up to 4 weeks for screening, treatment until clinically significant progression of disease, and 4 weeks of safety follow-up, and then long-term follow-up every 12 weeks.1 Cycle = 28 days.

DETAILED DESCRIPTION:
Up to 4 weeks for screening, treatment until clinically significant progression of disease, 4 weeks of safety follow-up and then long-term follow-up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants are included in the study if any of the following criteria apply:
* Participant is Black or African American, or American Indian or Alaska Native, or Native Hawaiian or Other Pacific Islander by self-identification.
* Previously received at least 2 and not more than 5 lines of systemic therapy for cGVHD.
* Receiving glucocorticoid therapy with a stable dose over the 2 weeks prior to screening.
* Have persistent cGVHD manifestations and systemic therapy is indicated.
* Karnofsky (if aged ≥ 16 years) / Lansky (if aged < 16 years) Performance Score of ≥ 60.
* At least 12 years of age; weight ≥ 40 kilograms (kg).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN).
* Total bilirubin ≤ 1.5 x ULN.
* Contraception (with double contraception methods) for male and female participants; not pregnant or breastfeeding for female participants
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* Participant has not been on a stable dose/regimen of systemic cGVHD treatment(s) for at least 2 weeks prior to screening. (Note: Concomitant corticosteroids, calcineurin inhibitors, sirolimus, MMF, methotrexate, rituximab, and ECP are acceptable. Systemic investigational GVHD treatments are not permitted).
* Histological relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
* Current treatment with ibrutinib or ruxolitinib. Prior treatment with ibrutinib or ruxolitinib is allowed with a washout of at least 28 days prior to enrollment.
* History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study (such as malabsorption syndromes, poorly controlled psychiatric disease, or coronary artery disease).
* Corrected QT interval using Fridericia's formula (QTc[F]) > 480 ms.
* Forced expiratory volume (in the first second; FEV1) ≤ 39% The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events and serious adverse events | Up to approximately 48 months
  Safety will be assessed by monitoring adverse events, physical Examinations, clinical laboratory evaluations, vital sign measurements, and ECG parameters.
Number of participants with clinically significant laboratory abnormalities | Up to approximately 12 months
Change from baseline in systolic and diastolic blood pressure | Baseline; up to approximately 12 months
Change from baseline in heart rate | Baseline; up to approximately 12 months
Change from baseline in corrected QT interval using Fridericia's formula (QTc[F]) | Baseline; up to approximately 12 months
Overall Response Rate (ORR) | Up to approximately 12 months
  The ORR is defined as the proportion of participants meeting the overall response criteria assessment of Complete Response (CR) or Partial Response (PR) as defined by the 2014 NIH Consensus Development Project on Clinical Trials in cGVHD at any post-baseline response assessment.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 12 months
  Assessments of DOR includes
  * The time from first response to progression, death, or new systemic therapy for cGVHD
  * Time from initial response to start of additional systemic cGVHD therapy or death
Change from baseline in the Lee Symptom Scale Score: Number of participants with a ≥ 7-point reduction | Baseline; up to approximately 12 months
  Changes in symptom burden/bother will be assessed using the Lee Symptom Scale, a symptom scale designed for individuals with chronic Graft Versus Host Disease (cGVHD). The questionnaire asks participants to indicate the degree of bother that they experienced due to symptoms in seven domains potentially affected by cGVHD (skin, eyes, mouth, breathing, eating and digestion, energy, and emotional distress). The response will be determined based on clinician's assessment.
Change from baseline in the Lee Symptom Scale Score: Number of participants with a ≥ 7-point reduction on 2 consecutive assessments | Baseline; up to approximately 12 months
  Changes in symptom burden/bother will be assessed using the Lee Symptom Scale, a symptom scale designed for individuals with chronic Graft Versus Host Disease (cGVHD). The questionnaire asks participants to indicate the degree of bother that they experienced due to symptoms in seven domains potentially affected by cGVHD (skin, eyes, mouth, breathing, eating and digestion, energy, and emotional distress). The response will be determined based on clinician's assessment.
Change from baseline in the Lee Symptom Scale Score: Duration of a ≥ 7 point reduction | Baseline; up to approximately 12 months
  Changes in symptom burden/bother will be assessed using the Lee Symptom Scale, a symptom scale designed for individuals with chronic Graft Versus Host Disease (cGVHD). The questionnaire asks participants to indicate the degree of bother that they experienced due to symptoms in seven domains potentially affected by cGVHD (skin, eyes, mouth, breathing, eating and digestion, energy, and emotional distress). The response will be determined based on clinician's assessment.
Response rate by organ system | Up to approximately 12 months
  The response rate for the nine individual organs (skin, eyes, mouth, esophagus, upper GI, lower GI, liver, lungs, and joints and fascia) will be assessed by the clinician.
Time to Response (TTR) | Up to approximately 12 months
  TTR defined as the time from the first dose of belumosudil to the first documented cGVHD response.
Time to Next Treatment (TTNT) | Up to approximately 12 months
  TTNT defined as the time from the first dose of belumosudil to the start of additional systemic cGVHD therapy.
Number of participants who have a best response of PR and CR | Up to approximately 12 months
  CR is defined as resolution of all manifestations of cGVHD in each organ or site. PR is defined as Improvement in at least 1 organ or site without progression in any other organ or site.
Change from baseline in corticosteroid dose | Baseline; up to approximately 12 months
  The prednisone equivalent dose of corticosteroids (mg/kg/day) during the study will be analyzed. The change in systemic corticosteroid dose over time will be determined.
Change from baseline in calcineurin inhibitor dose | Baseline; up to approximately 12 months
  The change in calcineurin inhibitor dose over time will be determined.
Failure-free survival (FFS) | Up to approximately 12 months
  FFS defined as the absence of new cGVHD systemic therapy, non-relapse mortality and recurrent malignancy. Median FFS (from first dose of belumosudil) will be analyzed.
Overall survival (OS) | Up to approximately 12 months
  OS defined as time from first dose of belumosudil to the date of death due to any cause.
Change from baseline in cGVHD global severity rating using the Clinician-Reported Global cGVHD Activity Assessment | Baseline; up to approximately 12 months
  Patient-reported outcome
Change from baseline in symptom activity as based on cGVHD Activity Assessment Patient Self-Report | Baseline; up to approximately 12 months
  Patient-reported outcome
Plasma belumosudil concentrations | Day 1 of Cycles 2, 3, 5, and 7 (1 Cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org